CLINICAL TRIAL: NCT03533179
Title: A Randomized, Participant-blinded Five-arm Crossover Study With Blinded Outcome Assessment Investigating Glucagon's Cardiovascular Effects With and Without Beta-blocker-induced Cardioinhibition.
Brief Title: Glucagon's Cardiovascular Effects With and Without Beta-blocker-induced Cardioinhibition
Acronym: GLUCAGON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Kasper Meidahl Petersen, MD, University Hospital Bispebjerg and Frederiksberg
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Glucagon+Beta-blocker
Record Dates: First submitted 2018-03-09; First posted 2018-05-23 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Drug Overdose; Overdose of Beta-adrenergic Blocking Drug
Keywords: Glucagon; Beta-adrenergic antagonist; poisoning
MeSH Terms: conditions — Drug Overdose; Poisoning | interventions — Glucagon; Glucagon-Like Peptide 1; esmolol; Saline Solution

STUDY DESIGN:
Intervention Model Description: 5-arm, participant and outcome-assessor blinded, randomized, placebo-controlled study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Interventions will be administered behind a curtain covering half the participant and thus the arm in which intervensions are administered. A list allocating participants to interventions are kept in an opaque envelope in a locked cabinet at the trial site. Outcome assessor will not have access to this list.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Esmolol-placebo+glucagon 1 placebo (A) (Experimental): Physiologic saline - esmolol dummy (10 mg esmolol/ml) is administered as a loading dose at baseline (time= -15 minutes) (corresponding to 0.125 ml/kg/min of saline). Continuous infusion (0.05-0.075 ml/kg/min) of saline is then administered until T=30 minutes.
  + Physiologic saline - glucagon dummy bolus 50 ml at time=0.
  Interventions: Drug: Physiologic saline - glucagon dummy; Drug: Physiologic saline - esmolol dummy
- Esmolol+glucagon 1 placebo (B) (Experimental): Esmolol intravenous solution (10 mg/ml esmolol hydrochloride) is administered as a loading dose (1.25 mg/kg/min esmolol) at baseline (time= -15 minutes). Continuous infusion (500-750 micrograms/kg/min) of esmolol/placebo is then administered until T=30 minutes.
  + Physiologic saline - glucagon dummy bolus (50 ml) at time=0.
  Interventions: Drug: Esmolol; Drug: Physiologic saline - glucagon dummy
- Esmolol+glucagon 1 (C) (Experimental): Esmolol intravenous solution (10 mg/ml esmolol hydrochloride) is administered as a loading dose (1.25 mg/kg/min esmolol) at baseline (time= -15 minutes). Continuous infusion (500-750 micrograms/kg/min) of esmolol/placebo is then administered until T=30 minutes.
  +Glukagon 1 (50 μg/kg bolus - over 1-3 min from time=0 min in 50 ml isotonic fluid)
  Interventions: Drug: Glucagon; Drug: Esmolol
- Esmolol-placebo+glucagon 2 (D) (Experimental): Physiologic saline - esmolol dummy (10 mg esmolol/ml) is administered as a loading dose at baseline (time= -15 minutes) (corresponding to 0.125 ml/kg/min of saline). Continuous infusion (0.05-0.075 ml/kg/min) of saline is then administered until T=30 minutes.
  +Glukagon 2 (50 μg/kg bolus - over 30 min in 50 ml isotonic fluid from time=0 min)
  Interventions: Drug: Glucagon; Drug: Physiologic saline - esmolol dummy
- Esmolol-placebo+glucagon 1 (E) (Experimental): Physiologic saline - esmolol dummy (10 mg esmolol/ml) is administered as a loading dose at baseline (time= -15 minutes) (corresponding to 0.125 ml/kg/min of saline). Continuous infusion (0.05-0.075 ml/kg/min) of saline is then administered until T=30 minutes.
  + Glukagon 1 (50 μg/kg bolus - over 1-3 min from time=0 min in 50 ml isotonic fluid)
  Interventions: Drug: Glucagon; Drug: Physiologic saline - esmolol dummy

INTERVENTIONS:
Drug: Glucagon — Glucagon 1 mg/ml solution is dissolved in 50 ml isotonic fluid and injected as bolus corresponding to 50 micrograms/kg over 1-3 minutes from time=0 on day C+E. on day D ("glucagon 2"), 50 micrograms/kg of glucagon is infused over 30 minutes from time=0 to time =30.
  Other Names: GlucaGen; ATC H04AA01
  Arms: Esmolol+glucagon 1 (C); Esmolol-placebo+glucagon 1 (E); Esmolol-placebo+glucagon 2 (D)
Drug: Esmolol — Esmolol hydrochloride 10 mg/ml is infused from time -15 min to time + 30 minutes as an initial bolus followed by an infusion. infusion rate is tapered if heart rate declines below 30 beats per minute (bpm) or >25 % from baseline, systolic blood pressure decreases below 80 mmHg or the participant experiences side effects.
  Other Names: Brevibloc; ATC C07AB09
  Arms: Esmolol+glucagon 1 (C); Esmolol+glucagon 1 placebo (B)
Drug: Physiologic saline - glucagon dummy — Isotonic 0.9 % sodium chloride solution is administered as matching placebo to glucagon, and injected in identical rates on corresponding days.
  Other Names: normal saline
  Arms: Esmolol+glucagon 1 placebo (B); Esmolol-placebo+glucagon 1 placebo (A)
Drug: Physiologic saline - esmolol dummy — Isotonic 0.9 % sodium chloride solution is administered as matching placebo to esmolol, and injected in identical rates on corresponding days.
  Other Names: normal saline
  Arms: Esmolol-placebo+glucagon 1 (E); Esmolol-placebo+glucagon 1 placebo (A); Esmolol-placebo+glucagon 2 (D)

SUMMARY:
This trial investigates effects of a glucagon bolus injection on heart rate, blood pressure and cardiac output during beta-blocker-induced cardiodepression. Furthermore, the effects of two different doses of intravenous glucagon on hemodynamic parameters are explored.

DETAILED DESCRIPTION:
This trial investigates effects of a glucagon bolus injection on heart rate, blood pressure and cardiac output during beta-blocker-induced cardiodepression. Furthermore, the effects of two different doses of intravenous glucagon on hemodynamic parameters are explored.

Glucagon, administered as a 50 micrograms/kg bolus injection which can be repeated or followed by continuous infusion (50 -150 micrograms / kg / hour) is a well-accepted and recommended treatment of beta-blocker poisoned patients [1-4]. The evidence for the recommended glucagon dose is based on animal trials and human case studies suggesting beneficial effects. Theoretically, high-dose glucagon mimics effect of beta-receptor agonists (increasing heart rate and cardiac output) [5] via activation of cardiac glucagon receptors, which cannot be blocked by beta blockers [1,6]. Glucagon receptors in the heart muscle are seemingly activated only at high glucagon levels [7] (but could also theoretically be an off-target effect); therefore the recommended glucagon dose for beta-blocker poisonings is higher than that recommended for reversal of hypoglycemia. Despite some animal and human case data suggesting beneficial effects of glucagon, other data suggest that glucagon may actually be inferior to other therapies of cardiovascular collapse due to cardioinhibitory drug poisonings [2]. It is important to keep in mind that the knowledge about glucagon's effects in poisoning situations is derived from uncontrolled cohort studies and case reports as well as animal studies [3,8]. Thus, the recommended dose has never been studied in a controlled clinical trial in humans. Therefore, the overall level of evidence pertaining to glucagon in the management of beta-blocker overdoses is low. There is a need for clinical human data investigating the glucagon doses recommended for treatment of beta-blocker overdose. The purpose of this participant- and outcome assessor blinded, randomized placebo-controlled crossover clinical trial is to investigate the effects of intravenous glucagon on the circulation alone or during beta-blocker-induced heart (rate) suppression. The trial includes a total of six visits; a screening visit and five trial days as described under Arms and Interventions. At the screening visit, anthropometric data (weight, height, blood pressure and pulse) is measured. Additionally, blood samples are collected in accordance with in/exclusion criteria. A spot urine sample measuring the albumin/creatinine ratio is collected and an electrocardiogram (ECG) is recorded to verify normality of heart rhythm and electrical impulses. In addition, an investigator carries out a clinical examination. Based on the clinical examination, urine and blood tests and ECG measurement, an investigator assesses whether the trial participant meet all inclusion criteria and no exclusion criteria. After screening and inclusion, participants will be invited to five trial days at the trial site (days A-E). The participant is blinded to interventions. On each day, participants are required to be fasting for 8±2 hours. A peripheral venous line is inserted into each antecubital vein. An arterial catheter connected to a pressure transducer is inserted into the radial artery in the wrist. In randomized order, one of the five interventions are performed (see below). A 5 lead ECG connected to a computer is placed on the participant. At T=-15 minutes, esmolol intravenous solution (10 mg esmolol/ml esmolol hydrochloride) or matching placebo is administered as a loading dose at baseline (time= -15 min) (corresponding to 1,25 mg/kg/min esmolol) [9]. Continuous infusion (500-750 micrograms/kg/min) of esmolol/placebo is then administered until T=30 minutes. Infusion is halted if heart rate decreases below 30 bpm or >25% from baseline, the systolic blood pressure drops below 80 mm Hg, or the participant experiences subjective side effects. Esmolol/placebo infusion stops at T=30 minutes. Glucagon (GlucaGen injectable solution) or saline solution is administered at time=0 minutes as an intravenous bolus (50 micrograms /kg over 1-2 minutes) on days C & E or as a continuous infusion (50 micrograms/kg over 30 min on day D). One point five grams of acetaminophen administered as a disintegrating tablet dissolved in 100 ml of water with guar gum is given orally shortly before study start on each day [10]. Repeated ECG's are recorded and blood is drawn for measurements of secondary biochemical endpoints. A drop of blood is used to test glucose levels using a blood glucose meter. Cardiovascular parameters (heart rate, blood pressure and pulse contour curve/arterial pressure wave) are recorded via the arterial catheter and pressure transducer connected to a computer. The participant is closely monitored on site until T=60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male determined by investigator, based upon physical examination, medical history, ECG, vital signs and laboratory results
* Body mass index (BMI) ≥ 18.5 and ≤ 29.9 kg/m2 and body weight between 50 and 100 kg, inclusive, at screening visit.

Exclusion Criteria:

* Abnormal blood levels of sodium, potassium, creatinine, alanine transaminase (ALT), alkaline phosphatase, albumin, bilirubin, hemoglobin, HbA1c, cholesterol fractions.
* Bradycardia (<45 beats per minute)
* Hypotension (systolic blood pressure < 100 mmHg)
* Second or third degree atrioventricular conduction delay
* Sick sinus syndrome
* Any heart disease or hypertension
* Pheochromocytoma
* Allergy to any active or inactive ingredient contained in investigatory medicines or tools.
* Raynaud's syndrome
* Prinzmetal's angina
* Diabetes
* Pulmonary disease
* Pheochromocytoma
* Any contraindication against investigatory medicines or tools.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male volunteers, determined healthy by medical history, physical examination including laboratory results
Enrollment: 10 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Heart rates on the esmolol+glucagon-day compared to the esmolol+placebo-day (2 minute average) | Glucagon bolus + 5±1 minute
  Arterial catheter connected to a pressure transducer records heart rate (beats per minute).

SECONDARY OUTCOMES:
Change in heart rate from baseline compared between study days. | -20, -10, 0, glucagon+3, +5, +10, +15, +20, +30, +40, +50, +60 minutes
  Arterial catheter connected to a pressure transducer records heart rate (beats per minute).
Change in stroke volume (ml) from baseline compared between study days. | -20, -10, 0, glucagon+3, +5, +10, +15, +20, +30, +40, +50, +60 minutes
  Stroke volume (ml) derived from arterial pulse contour analysis.
Change in systolic, diastolic and mean arterial pressure (mmHg) from baseline compared between study days. | -20, -10, 0, glucagon+3, +5, +10, +15, +20, +30, +40, +50, +60 minutes
  Arterial catheter connected to a pressure transducer records blood pressure in mm Hg.
Glucagon pharmacokinetics | Baseline and glucagon +2, +4, +6, +10, +15, +20, +30, +40, +50, +60 minutes
  Blood samples drawn for measurements of plasma glucagon
Effects of glucagon on blood glucose compared to placebo | Baseline and glucagon +2, +4, +6, +10, +15, +20, +30, +40, +50, +60 minutes
  Full blood glucose measured with a blood glucose meter
Adverse effects of glucagon | Baseline and glucagon +6,+10, +30, +60 minutes
  Nausea rated by a 4-point, verbal description scale (VDS) (no nausea=0, mild=1, moderate=2, severe=3).

OTHER OUTCOMES:
Effects of glucagon compared to placebo on gastric emptying time | Baseline and glucagon +10, +20, +30, +40, +50, +60 minutes
  Blood samples drawn for measurements of plasma paracetamol. Paracetamol is used as a tool for measuring gastric emptying time
Effects of glucagon compared to placebo on norepinephrine levels | T-20, T0, glucagon+5, +30, +60 minutes
  Blood samples drawn for measurements of norepinephrine.
Cardiac conductivity compared between days with glucagon1 and corresponding placebo days. | Baseline and glucagon +5, +10, +20, +30, +40, +50, +60 minutes
  5-lead ECG

CONTACTS AND LOCATIONS:
Overall Officials: Kasper M Petersen, MD, Principal Investigator — University Hospital Bispebjerg and Frederiksberg
Locations (1):
- University Hospital Bispebjerg, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brubacher JR. 62. β-adrenergic antagonists. In: Hoffman RS, Howland MA, Lewin NA, et al., eds. Goldfrank's toxicologic emergencies. New York: : McGraw-Hill Education 2015. 856-69.
- [Background] Graudins A, Lee HM, Druda D. Calcium channel antagonist and beta-blocker overdose: antidotes and adjunct therapies. Br J Clin Pharmacol. 2016 Mar;81(3):453-61. doi: 10.1111/bcp.12763. Epub 2015 Oct 30. PMID 26344579
- [Background] Bailey B. Glucagon in beta-blocker and calcium channel blocker overdoses: a systematic review. J Toxicol Clin Toxicol. 2003;41(5):595-602. doi: 10.1081/clt-120023761. PMID 14514004
- [Background] Beta blocker poisoning - UpToDate. https://www.uptodate.com/contents/beta-blocker-poisoning? search=beta%20blocker%20overdose&source=search_result&selectedTitle=1~14&usage_type=default&display_rank=1 (accessed 14 Feb 2018).
- [Background] Parmley WW, Glick G, Sonnenblick EH. Cardiovascular effects of glucagon in man. N Engl J Med. 1968 Jul 4;279(1):12-7. doi: 10.1056/NEJM196807042790103. No abstract available. PMID 4872564
- [Background] Yagami T. Differential coupling of glucagon and beta-adrenergic receptors with the small and large forms of the stimulatory G protein. Mol Pharmacol. 1995 Nov;48(5):849-54. PMID 7476915
- [Background] Rodgers RL. Glucagon and cyclic AMP: time to turn the page? Curr Diabetes Rev. 2012 Sep;8(5):362-81. doi: 10.2174/157339912802083540. PMID 22587514
- [Background] St-Onge M, Dube PA, Gosselin S, Guimont C, Godwin J, Archambault PM, Chauny JM, Frenette AJ, Darveau M, Le Sage N, Poitras J, Provencher J, Juurlink DN, Blais R. Treatment for calcium channel blocker poisoning: a systematic review. Clin Toxicol (Phila). 2014 Nov;52(9):926-44. doi: 10.3109/15563650.2014.965827. Epub 2014 Oct 6. PMID 25283255
- [Background] Reilly CS, Wood M, Koshakji RP, Wood AJ. Ultra-short-acting beta-blockade: a comparison with conventional beta-blockade. Clin Pharmacol Ther. 1985 Nov;38(5):579-85. doi: 10.1038/clpt.1985.227. PMID 2865029
- [Background] Medhus AW, Lofthus CM, Bredesen J, Husebye E. Gastric emptying: the validity of the paracetamol absorption test adjusted for individual pharmacokinetics. Neurogastroenterol Motil. 2001 Jun;13(3):179-85. doi: 10.1046/j.1365-2982.2001.00249.x. PMID 11437980
- [Derived] Petersen KM, Bogevig S, Riis T, Andersson NW, Dalhoff KP, Holst JJ, Knop FK, Faber J, Petersen TS, Christensen MB. High-Dose Glucagon Has Hemodynamic Effects Regardless of Cardiac Beta-Adrenoceptor Blockade: A Randomized Clinical Trial. J Am Heart Assoc. 2020 Nov 3;9(21):e016828. doi: 10.1161/JAHA.120.016828. Epub 2020 Oct 26. PMID 33103603

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT03533179/SAP_000.pdf